CLINICAL TRIAL: NCT00005862
Title: A Phase II Trial of SU5416 (NSC #696819) in Previously Treated Patients With Advanced, Metastatic and/or Locally Recurrent Soft Tissue Sarcomas
Brief Title: SU5416 in Treating Patients With Advanced, Metastatic, or Recurrent Soft Tissue Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067893; DFCI-00002; NCI-330
Record Dates: First submitted 2000-06-02; First posted 2004-02-12 (Estimated); Last update posted 2013-02-11 (Estimated); Status verified 2002-04

CONDITIONS: Gastrointestinal Stromal Tumor; Sarcoma
Keywords: stage III adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; gastrointestinal stromal tumor; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Sarcoma | interventions — Semaxinib

ARMS (1):
- Arm I (Experimental): atients receive SU5416 IV twice weekly for 4 weeks. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: semaxanib

INTERVENTIONS:
Drug: semaxanib

SUMMARY:
Phase II trial to study the effectiveness of SU5416 in treating patients who have advanced, metastatic, or recurrent soft tissue sarcomas. SU5416 may stop the growth of soft tissue sarcomas by stopping blood flow to the tumor.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate, response duration, and overall survival in patients with advanced, metastatic, or recurrent soft tissue sarcoma or gastrointestinal stromal tumor when treated with SU5416.

II. Determine the safety of SU5416 in these patients.

OUTLINE: This is a multicenter study.

Patients receive SU5416 IV twice weekly for 4 weeks. Treatment continues every 4 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly for 3 months and then every 3 months for 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed advanced, metastatic, recurrent, or unresectable soft tissue sarcoma or gastrointestinal stromal tumor
* Measurable disease defined as lesions that can be measured in at least one dimension as at least 20 mm with conventional techniques or at least 10 mm with spiral CT scan
* Must have received prior chemotherapy with no response or progression after initial response
* Evidence of disease progression in past 3 months
* No CNS metastases or primary brain tumors

PATIENT CHARACTERISTICS:

* Age: 18 and over
* Performance status: ECOG 0-1
* Life expectancy: At least 12 weeks
* WBC greater than 2,000/mm3
* Platelet count greater than 100,000/mm3
* Fibrin split products no greater than 0.001 mg
* Fibrinogen greater than 200 mg/dL
* Bilirubin no greater than upper limit of normal (ULN)
* AST/ALT less than 1.5 times ULN
* PT/PTT less than 1.25 times ULN
* Creatinine no greater than 1.5 mg/dL
* At least 1 year since bypass surgery for atherosclerotic coronary artery disease
* No uncompensated coronary artery disease
* No history of myocardial infarction or unstable/severe angina in past 6 months
* No severe peripheral vascular disease
* No history of deep venous or arterial thrombosis in past 3 months
* No history of pulmonary embolism in past 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No diabetes mellitus
* No history of bleeding diathesis
* No known active retroviral disease
* No AIDS-associated Kaposi's sarcoma
* No history of allergic reaction to Cremophor or paclitaxel
* No uncontrolled illness or psychiatric disorder that would preclude study

PRIOR CONCURRENT THERAPY:

* No concurrent immunotherapy
* At least 3 weeks since prior chemotherapy (6 weeks since mitomycin or nitrosoureas)
* No concurrent chemotherapy
* At least 3 weeks since prior radiotherapy
* No concurrent radiotherapy
* Greater than 2 weeks since prior minor surgery (greater than 4 weeks since major surgery)
* No concurrent antiinflammatory drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2000-10; Primary Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George D. Demetri, MD, Study Chair — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts